CLINICAL TRIAL: NCT03578926
Title: Performance of Toric Silicone Hydrogel Contact Lenses Following Two Weeks of Daily Wear
Brief Title: Performance of Two Toric Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-93
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double masked, bilateral, 2-weeks, crossover study.
Who Masked: Participant, Investigator
Masking Description: Double masked (participant and investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- fanfilcon A toric lens (Experimental): Randomized participants will wear fanfilcon A toric contact lenses bilaterally for two weeks then switch to senofilcon A toric contact lenses for another two weeks.
  Interventions: Device: fanfilcon A toric lens
- senofilcon A toric lens (Active Comparator): Randomized participants will wear senofilcon A toric contact lenses bilaterally for two weeks then switch to fanfilcon A toric contact lenses for another two weeks.
  Interventions: Device: senofilcon A toric lens

INTERVENTIONS:
Device: fanfilcon A toric lens — contact lens
  Other Names: Avaira Vitality toric lens
  Arms: fanfilcon A toric lens
Device: senofilcon A toric lens — contact lens
  Other Names: Acuvue Oasys for Astigmatism
  Arms: senofilcon A toric lens

SUMMARY:
Prospective study to evaluate the clinical performance of fanfilcon A toric contact lens and senofilcon A toric contact lens after two weeks of wear.

DETAILED DESCRIPTION:
The aim of this prospective study is to evaluate the clinical performance of Avaira Vitality toric and ACUVUE OASYS® for ASTIGMATISM contact lenses after 2-weeks of wear in each pair.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted soft contact lens wearer
* Has a contact lens spherical prescription between +6.00 to - 9.00 (inclusive)
* Have no less than -0.75D of astigmatism and no more than -2.25 D in both eyes.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter.
* Patient contact lens refraction should fit within the available parameters of the study lenses.
* Is willing to comply with the wear schedule (at least 5 days per week, > 8 hours/day assuming there are no contraindications for doing so).
* Is willing to comply with the visit schedule

Exclusion Criteria:

* Has a CL prescription outside the range of the available parameters of the study lenses.
* Has a spectacle cylinder less than -0.75D or more than -2.50 D of cylinder in either eye.
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
* Presence of clinically significant (grade 2-4) anterior segment abnormalities
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as:
* Pathological dry eye or associated findings
* Pterygium, pinguecula, or corneal scars within the visual axis
* Neovascularization > 0.75 mm in from of the limbus
* Giant papillary conjunctivitis (GCP) worse than grade 1
* Anterior uveitis or iritis (past or present)
* Seborrheic eczema, Seborrheic conjunctivitis
* History of corneal ulcers or fungal infections
* Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Velázquez Guerrero, MSc., FIACLE, Principal Investigator — School of Optometry, National Autonomous University
Locations (1):
- Optometry Clinic, National Autonomous University, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 45 habitual lens wearers were enrolled. 1 participant was ineligible for the study due to an unacceptable lens fit. 44 participants were dispensed and completed all study visits.
Groups:
- Fanfilcon A Toric: Randomized participants will wear fanfilcon A toric contact lenses bilaterally for two weeks then switch to senofilcon A toric contact lenses for another two weeks.
  Contact Lens: fanfilcon A toric
- Senofilcon A Toric: Randomized participants will wear senofilcon A toric contact lenses bilaterally for two weeks then switch to fanfilcon A toric contact lenses for another two weeks.
  Contact Lens: senofilcon A toric
Period: First Intervention
Arm/Group | Fanfilcon A Toric | Senofilcon A Toric
Started | 21 | 23
Completed | 21 | 23
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Fanfilcon A Toric | Senofilcon A Toric
Started | 23 | 21
Completed | 23 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 45 subjects were enrolled. One participant was ineligible for the study due to an unacceptable lens fit at the first visit. A total of 44 subjects were dispensed and completed all study visits.
Groups:
- Overall Study: All subjects are randomized to 2-week cross-over study to compare fanfilcon A and senofilcon A.
Arm/Group | Overall Study
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 44

OUTCOME MEASURES:

1. Primary Outcome: Lens Centration
Description: Centration of lens on eye (Optimum, Decentration acceptable, Decentration unacceptable)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Fanfilcon A: Randomized participants will wear fanfilcon A toric contact lenses bilaterally for two weeks then switch to senofilcon A toric contact lenses for another two weeks.
  contact lens: fanfilcon A
- Senofilcon A: Randomized participants will wear senofilcon A toric contact lenses bilaterally for two weeks then switch to fanfilcon A toric contact lenses for another two weeks.
  contact lens: senofilcon A
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 44 | 44
Participants | 44 | 44

2. Primary Outcome: Lens Centration
Description: Centration of lens on eye (Optimum, Decentration acceptable, Decentration unacceptable)
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 44 | 44
Participants
  Optimal Centration | 44 | 44
  Decentration Acceptable | 0 | 0
  Decentration unacceptable | 0 | 0

3. Primary Outcome: Corneal Coverage
Description: Lens covering the cornea (Yes, No)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 44 | 44
Participants
  Yes | 44 | 44
  No | 0 | 0

4. Primary Outcome: Corneal Coverage
Description: Lens covering the cornea (Yes, No)
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 44 | 44
Participants
  Yes | 44 | 44
  No | 0 | 0

5. Primary Outcome: Post Blink Movement
Description: Amount of lens movement after blink (0-5 Likert Scale, 0=Insufficient, 2=Optimal, 4=Excessive movement)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 44 | 44
units on a scale | 1.91 (0.3) | 1.98 (0.3)

6. Primary Outcome: Post Blink Movement
Description: Amount of lens movement after blink (0-5 Likert Scale, 0=Insufficient, 2=Optimal, 4=Excessive movement)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A | Senofilcon A
Number analyzed (Participants) | 44 | 44
units on a scale | 2.00 (0.0) | 2.02 (0.3)

7. Secondary Outcome: Wearing Time
Description: Average daily wearing time (hours/day)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Groups:
- Fanfilcon A - 2 Weeks: Randomized participants will wear fanfilcon A toric contact lenses bilaterally for two weeks then switch to senofilcon A toric contact lenses for another two weeks.
  fanfilcon A: contact lens
- Senofilcon A - 2 Weeks: Randomized participants will wear senofilcon A toric contact lenses bilaterally for two weeks then switch to fanfilcon A toric contact lenses for another two weeks.
  senofilcon A: contact lens
Arm/Group | Fanfilcon A - 2 Weeks | Senofilcon A - 2 Weeks
Number analyzed (Participants) | 44 | 44
hours/day | 12.2 (2.9) | 11.6 (3.1)

8. Secondary Outcome: Comfortable Wearing Time
Description: Comfortable daily wearing time (hours/day)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Fanfilcon A - 2 Weeks | Senofilcon A - 2 Weeks
Number analyzed (Participants) | 44 | 44
hours/day | 10.0 (3.2) | 9.0 (3.0)

ADVERSE EVENTS:
Time Frame: 2 weeks during each crossover period
Groups:
- Fanfilcon A: Randomized participants will wear fanfilcon A toric contact lenses bilaterally for two weeks then switch to senofilcon A toric contact lenses for another two weeks.
  fanfilcon A toric lens: contact lens
- Senofilcon A: Randomized participants will wear senofilcon A toric contact lenses bilaterally for two weeks then switch to fanfilcon A toric contact lenses for another two weeks.
  senofilcon A toric lens: contact lens
Arm/Group | Fanfilcon A | Senofilcon A
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT03578926/Prot_SAP_000.pdf